CLINICAL TRIAL: NCT06997172
Title: Determining the Short- to Medium-term Outcome After Minimally Invasive Sonography Guided Release of the Carpal Tunnel Compared to Standard-of-care Open and Endoscopic Techniques: a Randomized Controlled Superiority Trial With an Internal Pilot-phase
Brief Title: Short- to Medium-term Outcome of Minimally Invasive Carpal Tunnel Release
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-00406; mu25Kamphuis
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Carpal Tunnel
Keywords: Percutaneous sonography guided release
MeSH Terms: conditions — Median Neuropathy | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TCTR (thread carpal tunnel release) (Experimental): Percutaneous sonography guided release of carpal tunnel
  Interventions: Procedure: TCTR (thread carpal tunnel release)
- Standard of care technique (Active Comparator): Standard of care technique (consisting of either the open or endoscopic technique) release of carpal tunnel
  Interventions: Procedure: Standard-of-care

INTERVENTIONS:
Procedure: TCTR (thread carpal tunnel release) — Percutaneous sonography guided release of carpal tunnel release
  Arms: TCTR (thread carpal tunnel release)
Procedure: Standard-of-care — Open or endoscopic carpal tunnel release based on patients' and physicians' preferences
  Arms: Standard of care technique

SUMMARY:
The aim of the study is to determine whether minimally invasive, ultrasound-guided thread carpal tunnel release leads to faster functional recovery compared to standard open and endoscopic techniques in patients with carpal tunnel syndrome.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is the most common peripheral nerve compression disorder encountered in hand surgery. It affects a broad demographic, from young women (often linked to pregnancy and breastfeeding) and young men involved in manual labor, to elderly individuals. The condition causes pain, numbness, and functional impairment in the hand, which can progress to permanent disability if untreated. Typically, conservative treatment (e.g., night splints, corticosteroid injections) is the first step. However, when symptoms persist, surgical decompression of the median nerve becomes necessary.

The current gold standard for surgical treatment of CTS is open carpal tunnel release (OCTR). This involves making a 2-5 cm incision in the palm and cutting the transverse carpal ligament under direct vision. While effective in relieving nerve compression, this approach creates a scar in the load-bearing area of the palm, which can lead to prolonged post-operative pain, delayed wound healing, reduced grip strength, extended rehabilitation time and limitations in early hand use.

To address some of these drawbacks, endoscopic carpal tunnel release (ECTR) was developed. This technique uses a smaller incision at the wrist and a camera system to visualize and divide the ligament. While less invasive than OCTR, ECTR still involves an incision, and significant scar tissue may still develop, especially internally.

Both techniques require postoperative wound care, stitch removal, and carry risks of complications such as nerve or tendon injury, infection, or incomplete release. Additionally, these methods often result in delays in returning to work and daily activities, particularly burdensome for patients in physically demanding jobs.

In recent years, a novel percutaneous ultrasound-guided technique, known as thread carpal tunnel release (TCTR), has been introduced. This method uses two small puncture sites instead of incisions. Under real-time ultrasound guidance, a suture loop is passed around the transverse carpal ligament, which is then divided using a sawing motion. This technique bears several advantages including absence of external scar, reduced postoperative pain, no requirement for stitch removal, potential faster recovery allowing earlier return to normal function, daily activities and work.

The theoretical benefits of TCTR are supported by cadaveric and small clinical studies, but no large randomized controlled trials have yet compared TCTR directly with both open and endoscopic techniques. This study aims to fill that evidence gap by rigorously evaluating whether TCTR leads to quicker functional recovery, measured via validated functional assessments in a real-world clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older
* Electroneurographically proven carpal tunnel syndrome
* Informed Consent for trial participation

Exclusion Criteria:

* Revision surgery
* Inability to give informed consent, whether it be due to an insurmountable language barrier or another reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
The objective functional assessment of the BCTQ score at 2 weeks | 2 weeks post-operative
  Functional assessment of the BCTQ. The BCTQ is a patient reported outcome measure (PROM) questionnaire that examines subjective symptom severity and objective overall functional status. The Functional Status Scale evaluates the ability of the patient to use their hand in daily life using 8 questions, which are scored from 1-5 with 1 as no difficulty and 5 as difficult. Therefore, the higher the score, the more difficulty the patient has with the symptom.

SECONDARY OUTCOMES:
The objective functional assessment of the BCTQ score | 4 and 6 weeks and 6 month post-operative
  Functional assessment of the BCTQ. The BCTQ is a patient reported outcome measure (PROM) questionnaire that examines subjective symptom severity and objective overall functional status. The Functional Status Scale evaluates the ability of the patient to use their hand in daily life using 8 questions, which are scored from 1-5 with 1 as no difficulty and 5 as difficult. Therefore, the higher the score, the more difficulty the patient has with the symptom
Overall BCTQ score, which is a combination of the subjective symptom severity and the objective functional status. | 2, 4 and 6 weeks and 6 months post-operative
  The BCTQ is a patient reported outcome measure (PROM) questionnaire that examines subjective symptom severity and objective overall functional status. The Symptom Severity Scale with 11 questions is scored on a Likert scale of 1-5 and the Functional Status Scale with 8 questions is scored from 1-5 with 1 as no difficulty and 5 as difficult. Therefore, the higher the score, the more difficulty the patient has with the symptom.
The subjective symptom severity score of the BCTQ | 2, 4 and 6 weeks and 6 months post-operative
  The BCTQ is a patient reported outcome measure (PROM) questionnaire that examines subjective symptom severity and objective overall functional status. The Symptom Severity Scale describes the symptoms concerning sensibility and pain and is evaluated using 11 questions scored on a Likert scale of 1-5 with 1 as no difficulty and 5 as difficult. Therefore, the higher the score, the more difficulty the patient has with the symptom.
Hand-specific health | 2, 4 and 6 weeks and 6 months post-operative
  The Michigan Hand Questionnaire (MHQ)is one of the most widely utilized, hand-specific surveys that measures health status relevant to patients with acute and chronic hand disorders.Scale ranges from 0-100, while lower scores indicate better outcomes.
Functional recovery time | up to 6 months post-operative
  Days until return to daily activities and/or work
Recovery from pain | up to 6 months post-operative
  Days until discontinuation of pain medication
Area of the median nerve | 2, 4 and 6 weeks and 6 months post-operative
  Cross sectional area of the median nerve (cm2) is investigatad by sonographic
Range of motion | 2, 4 and 6 weeks and 6 months post-operative
  Range of motion in degrees
thenar atrophies | 2, 4 and 6 weeks and 6 months post-operative
  Presence of thenar atrophies (yes / no)
Strength in the abductor pollicis brevis | 2, 4 and 6 weeks and 6 months post-operative
  Force Abductor pollicis brevis in Medical Research Council (MCR) grade. The force produced by the abductor pollicis brevis (APB) muscle is graded using the Medical Research Council (MRC) scale, which assesses muscle strength, ranging vrom 0-5. A grade 5 indicates full strength and normal function, while lower grades indicate varying degrees of weakness.
Two-point discrimination | 2, 4 and 6 weeks and 6 months post-operative
  two-point discrimination in millimeter
Grip strength | 2, 4 and 6 weeks and 6 months post-operative
  Grip strength is measured with the Jamar dynamometer
Pinch strength | 2, 4 and 6 weeks and 6 months post-operative
  Pinch strength is measured with the Jamar dynamometer
Pain intensity | 2, 4 and 6 weeks and 6 months post-operative
  Pain measured with the visual analog scale (VAS) from 0-10
Outcome satisfaction | 2, 4 and 6 weeks and 6 months post-operative
  Patient satisfaction measured with the VAS from 0-10

CONTACTS AND LOCATIONS:
Overall Officials: Saskia Kamphuis, Study Chair — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland